CLINICAL TRIAL: NCT05886972
Title: Effect Of Patient Awareness About Possibility Of Occurrence Of Pain During Propofol Injection On The Rate Of Incidence And Severity Of Pain During Injection ; A Randomized Controlled Study.
Brief Title: Effect Of Patient Awareness About Possibility Of Occurrence Of Pain During Propofol Injection On The Rate Of Incidence And Severity Of Pain During Injection .
Acronym: No acronym
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahmoud Hussein Bahr, Associated Professor of Anesthesiology and Surgical Intensive Care and pain medicine, Beni-Suef University
Other Study IDs: FMBSUREC/02052023/sayem
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Effect of Patient Awareness on Incidence and Severity of Propofol Injection Induced Pain
Keywords: Propofol injection induced pain; Patient awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients aware about propofol injection induced pain: Patients who will be informed about the possibility of incidence of propofol injection pain
  Interventions: Behavioral: Awareness about propofol injection induced pain
- Patients not aware about propofol injection induced pain: Patients will not be informed about the possibility of incidence of propofol injection pain
  Interventions: Behavioral: Awareness about propofol injection induced pain

INTERVENTIONS:
Behavioral: Awareness about propofol injection induced pain — The aim of the study is to observe the effect of patient awareness about the possibility of occurrence of pain during propofol injection on the rate of incidence and severity of pain during injection as a primary goal as the pain score of propofol injection pain is the main end point of the study .

SUMMARY:
Propofol is the most common intravenous (IV) anesthetic agent, used for anesthesia induction and maintenance during surgeries due to its rapid onset and short duration.

However, the incidence of propofol injection pain occurs in about 20% to 90% of patients that can decrease patient satisfaction and safety .

Awareness of patient about propofol injection pain can affect patient anxiety and stress that will be reflected on incidence and severity of occurance of propofol injection pain. In our study the effect of patient awareness on propofol injection pain will be evaluated after adequate using of the pharmacological and non-pharmacological therapy that have been demonstrated to be effective in attenuating injection pain.

DETAILED DESCRIPTION:
Propofol is the most common intravenous (IV) anesthetic agent, used for anesthesia induction and maintenance during surgeries due to its rapid onset and short duration .

However, the incidence of propofol injection pain occurs in about 20% to 90% of patients that can decrease patient satisfaction and safety .

The mechanism of propofol injection pain has not been known yet, but many factors are involved that include the intrinsic drug property (e.g. emulsion composition, pH of the formulation, temperature, injection volume and osmolarity) .

As the lipid solvent irritates the venous intima and triggers a local kallikrein kinin cascade by discharging bradykinin and inflammatory factors, and injection pain occurs when peripheral nerve endings are directly exposed to propofol .

Other factors, including the site of injection, speed of injection, vein size, blood buffering, sex and simultaneous use of different drugs, seem to affect the incidence and severity of propofol injection pain .

The incidence and the severity of pain following propofol injection is increased in peripheral site of injection , smaller size of the vessels and slow injection and the pain can be reduced by rapid injection of propofol into the large sized veins as veins of antecubital fossa, however, this is not always practical in clinical practice .

Propofol injection pain is more common and more sever in females than males and the suggested reason of gender difference is due to the mechanical effect that male has a larger venous size than female while another factor suggested is the difference of pain sensitivity observed between the gender.

Low education level also increases the incidence and the severity of propofol injection pain as high education level will help during the patients' preoperative preparations and will reduce preoperative anxiety .

Psychogenic factors such as anxiety, depression, and fear of pain are frequently observed in patients undergoing elective surgery. Among these, preoperative anxiety and pain sensitivity has been the most important factors .

Preoperative anxiety activates the release of neuroendocrine mediators related to stress response and negatively affects anesthetic methods, surgical recovery, and postoperative pain levels .

Awareness of patient about propofol injection pain can affect patient anxiety and stress that will be reflected on incidence and severity of occurance of propofol injection pain. In our study the effect of patient awareness on propofol injection pain will be evaluated after adequate using of the pharmacological and non-pharmacological therapy that have been demonstrated to be effective in attenuating injection pain.

Many approaches have been recommended to decrease propofol injection pain including both pharmacological (e.g. pre-treatment with Paracetamol , lidocaine, magnesium sulfate, ketamine , ondansetron , Granisetron ,and and triglycerides ) .

It is generally approved that lidocaine is an adequate anesthetic that precludes injection pain. However, its adverse cardiovascular and hemodynamic effects and swelling at its injection site require to be further studied .

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 20 to 40 years of The American Society of Anesthesiologists (ASA) I-II , who will be undergoing elective surgery under general anesthesia

Exclusion Criteria:

* patient with mental illness, poor understanding or difficulty in communication or pain assessment .
* any organ dysfunction, neurological disease, diabetes mellitus .
* patient with high education level (patient with education level after high secondary school) .
* patient with Body Mass Index (BMI) < 18 or > 30
* allergy to the study drugs .
* history of chronic pain or those taking regular analgesics, anti-inflammatory drugs pre-operatively .

history of drug abuse and other contraindication for lidocaine such as severe bradycardia, Wolf-Parkinson-White syndrome, and other tachyarrhythmias .

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pain threshold is different between males and females , so the study needs one gender
Study Population: the study will be performed on 210 patients , 2 equal groups. Group A (Aware group): who will be informed about the possibility of incidence of propofol injection pain Group B ( Un aware group) : who will not be informed about the possibility of incidence of propofol injection pain
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment | During first 10 seconds after receiving first dose of propofol
  Pain intensity will be measured by Verbal categorical scoring (VCS) Verbal categorical scoring (VCS) is a 4-point pain scale: 0-no pain, 1-mild pain with no behavioral sign, 2-moderate pain accompanied by a behavioral sign, and 3-severe pain with a strong vocal response accompanied by facial grimacing, arm withdrawal, or crying ( Jeon Y ,2012).

SECONDARY OUTCOMES:
Age | Preoperative visit
  Age per years
Weight | Preoperative visit
  Weight by kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Hussein Bahr, Beni-suef, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet